CLINICAL TRIAL: NCT05877937
Title: Effect of Humor on Pain and Anxiety in Patients With Rheumatoid Arthritis: A Prospective, Randomized Controlled Study
Brief Title: Humor Therapy and Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Güler Balci Alparslan, Prof. Dr., Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202042005
Record Dates: First submitted 2023-03-02; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Pain; Anxiety; Rheumatoid Arthritis; Nursing Caries
MeSH Terms: conditions — Pain; Anxiety Disorders; Arthritis, Rheumatoid | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventions group (Experimental): The intervention group watched a comedy movie during routine IV biologic treatment in the chemotherapy day unit.
  Interventions: Other: Supportive care (Watching a comedy movie)
- Control group (No Intervention): The control group received only routine IV biologic treatment as a usual care.

INTERVENTIONS:
Other: Supportive care (Watching a comedy movie) — A 10.1 inch Android tablet (2 pieces) and disposable earplugs for each patient were used in the study. A comic film archive was created in line with the recommendation and consultancy of department of state conservatory and performing arts. In this regard, the officials of the Conservatory stated that they had no standardized comedy films specific to society and emphasized that the standardization of art limits art activities. Therefore, there should be no limitations for art. In the film archive cre-ated according to their suggestions, there were a total of five comedy movies, including three Turkish comedies, one foreign romantic comedy, and one foreign Turkish-dubbed family comedy. The original/licensed versions of the movies in this archive were ob-tained and uploaded to the tablet. The movies lasted 90-120 minutes (as long as the av-erage duration of IV treatment). The patients selected the movie that they would watch during the treatment.
  Arms: Interventions group

SUMMARY:
The goal of this prospective, randomized controlled study was to inverstigate the effect of humor on pain and in patients with rheumatoid arthritis (RA) during IV treatment. The main question[s] it aims to answer are:

* to compare the effect of humor on pain between two groups of patients with RA who watched a comedy movie (intervention group) and who did not (control group) during IV biological therapy.
* to compare the effect of humor on anxiety between two groups of patients with RA who watched a comedy movie (intervention group) and who did not (control group) during IV biological therapy.

Participants in the intervention group watched a comedy movie during routine IV biologic treatment in the chemotherapy unit, while the control group received only routine IV biologic treatment as a usual care.

DETAILED DESCRIPTION:
Settings and Participants This study included a total of 36 patients who were diagnosed with RA according to the criteria of the American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) (Aletaha et al. 2010) and received IV biological drug therapy in the chemotherapy day unit of an oncology clinic between September 2020 and November 2021. In addition to hematological and oncological patients receiving outpatient chemotherapy, patients receiving outpatient IV/subcutaneous biologic drug therapy were also treated in the chemotherapy day unit. As a result of the posterior power analysis, the power was calculated as 1.00 (100%) for the VAS with n=36. The patients were randomized allocated two groups: Intervention group and control group. Both groups received routine IV biologic treatment.The allocation ratio was set 1:1.

Inclusion criteria The following study inclusion criteria were used: having reached the age of 18; having been given a diagnosis of RA in accordance with the ACR/EULAR (9) classification criteria at least six months prior to the study; receiving IV biologic infusion therapy in the chemotherapy day unit; not having any other inflammatory diseases; experiencing pain that ranged from 4 to 8 on the VAS; not having been given a complex disease, such as cancer; not being pregnant; and having no mental diagnosis, no drug use-related or disease-related impairment of consciousness, no communication issue, and voluntary participation in the study.

Exclusion criteria The exclusion criteria were the following: a switch in treatment method during the intervention or any discomfort such as dizziness or nausea while watching a comic film.

Outcomes were assessed as pre-post test immediately before and after the IV biologic infusion treatment:

* Pre-test: Before the IV infusion treatment, the patients were evaluated face-to-face by the researcher in an empty quiet examination room in the chemotherapy day unit using a descriptive information form, the Visual Analog Scale (VAS), and the State-Trait Anxiety Inventory (STAI).
* Post-test: After the IV infusion treatment (post-test), the patients were re-evaluated using the VAS and the SAI.

ELIGIBILITY:
Inclusion Criteria:

* having reached the age of 18; having been given a diagnosis of RA in accordance with the ACR/EULAR (Aletaha et al. 2010) classification criteria at least six months prior to the study; receiving IV biologic infusion therapy in the chemotherapy day unit; not having any other inflammatory diseases; experiencing pain that ranged from 4 to 8 on the VAS; not having been given a complex disease, such as cancer; not being pregnant; and having no mental diagnosis, no drug use-related or disease-related impairment of consciousness, no communication issue, and voluntary participation in the study.

Exclusion Criteria:

* a switch in treatment method during the intervention or any discomfort such as dizzi-ness or nausea while watching a comic film.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | VAS score will evaluate at baseline (immediately before the IV biologic infusion treatment)
  VAS is the pain rating scale. A VAS consists of a line, often 10 cm long, with verbal anchors at either end, similar to an NRS (e.g., "no pain" on the far left and "the most intense pain imaginable" on the far right). The patient places a mark at a point on the line corresponding to the patient's rating of pain intensity.
Visual Analog Scale (VAS) | VAS score will evaluate direct after the IV biologic infusion treatment
  VAS is the pain rating scale. A VAS consists of a line, often 10 cm long, with verbal anchors at either end, similar to an NRS (e.g., "no pain" on the far left and "the most intense pain imaginable" on the far right). The patient places a mark at a point on the line corresponding to the patient's rating of pain intensity.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | STAI scores will evaluate at baseline (immediatley before the IV biologic infusion treatment)
  The State-Trait Anxiety Inventory was developed in 1970 and adapted to Turkish in 1977 (11,12). This is a four-point Likert-type scale with two parts, where the first and second parts include questions to determine one's state and trait anxiety levels, respectively. Our study used the first part, called the State Anxiety Scale. The total scale score varies between 20 and 80. A higher score indicates higher anxiety. The Cronbach's alpha is 0.82 for the STAI.
State-Trait Anxiety Inventory (STAI) | STAI scores will evaluate direkt after the IV biologic infusion treatment.
  The State-Trait Anxiety Inventory was developed in 1970 and adapted to Turkish in 1977 (11,12). This is a four-point Likert-type scale with two parts, where the first and second parts include questions to determine one's state and trait anxiety levels, respectively. Our study used the first part, called the State Anxiety Scale. The total scale score varies between 20 and 80. A higher score indicates higher anxiety. The Cronbach's alpha is 0.82 for the STAI.

CONTACTS AND LOCATIONS:
Overall Officials: Güler Balci Alparslan, Study Director — Eskisehir Osmangazi University, Faculty of Health Science, Department of Internal Medicine Nursing
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No